CLINICAL TRIAL: NCT01735695
Title: Performance Evaluation Study for a New Meconium Detection Test
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Laniado Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Laniado25112012; Laniado25122012-1 (Other: Laniado Hospital)
Record Dates: First submitted 2012-11-25; First posted 2012-11-28 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Pregnancy
Keywords: Meconium; concentration; level

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to collect amniotic fluid samples from pregnant women. Amniotic fluid samples will be tested for meconium with a new assay. The results will be correlated with other laboratory tests.

DETAILED DESCRIPTION:
Female volunteers will be recruited locally in a single medical center. After the occurrence of amniotic membranes rupture, amniotic fluid samples will be collected extracorporeally.

Meconium concentration levels will be measured by the new test. Other laboratory tests will be employed in order to determine the accuracy of the new test.

ELIGIBILITY:
Inclusion Criteria:

* Provide written or oral informed consent to participate in the study and agree to comply with study procedures.
* Pregnant.
* Intend to seek medical care during pregnancy.

Exclusion Criteria:

* Amniotic fluid samples are mixed with urine.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-08 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Meconium concentration in amniotic fluid | One year

CONTACTS AND LOCATIONS:
Overall Officials: Brigita Wintrov, MD, Study Director — Laniado Medical Center
Locations (1):
- Laniado Hospital, Netanya, Israel